CLINICAL TRIAL: NCT06814457
Title: The Effect of Nursing Care Bundle on Oral Intake Among Critically Ill Children With Post-Extubation Dysphagia: Randomized Control Study
Brief Title: Nursing Care Bundle on Oral Intake Among Critically Ill Children With Post-Extubation Dysphagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Eman Wardany Abdelaal Mohamed, assistant professor of pediatric nursing, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KafrelsheikhU5
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Oropharyngeal Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional care group (No Intervention): Consisted of 30 children who will receive conventional hospital care with no additional interventions.
- Care bundle group (Experimental): Consisted of 30 children who will receive a nursing care bundle for enhancing oral intake
  Interventions: Procedure: a nursing care bundle on oral intake

INTERVENTIONS:
Procedure: a nursing care bundle on oral intake — a nursing care bundle on oral intake will be started the day after their successful extubation and extend for 14th days. Additionally, the participants will be provided with a brief education on safe swallowing.
  Arms: Care bundle group

SUMMARY:
the aim of this study is to evaluate the effect of Nursing care Bundle on Oral Intake among Critically Ill Children with Post-Extubation Dysphagia

DETAILED DESCRIPTION:
The researchers explained the study's aim, benefits, and procedures for participation, after that the parents of the children provided an informed consent. children's baseline data was collected from their records prior to intervention in order to identify children who meet the required criteria of the study. then the participants were selected and divided randomly (using a simple random method) into two equal groups. One subject for the control group, one for the study group, and so on, distributed the participants into two equivalent groups as fellow:

Control Group: Consisted of 30 children who will receive conventional hospital care with no additional interventions.

Study Group: Consisted of 30 children who will receive a nursing care bundle on oral intake starting the day after their successful extubation and extend for 14th days. Additionally, the participants were provided with a brief education on safe swallowing.

ELIGIBILITY:
Inclusion Criteria:

* undergoing emergency oral endotracheal intubation for at least 48 hours
* able to communicate and having no sensory deficit and accepted to participate in the research

Exclusion Criteria:

* children who had a history of neuromuscular disease, preexisting swallowing problems and agitated children were excluded.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of oral health post-extubation on Post-Extubation Oral Assessment Scale | The first measurement time will be From extubation of mechanical ventilation up to 1 week"7 th day's post-extubation". The second time will be from extubation up to 2 week"14th day's" post-extubation
  It consisted of eight categories including Voice, ability to swallow, lips, saliva, tongue, mucous membranes, gingiva and teeth. scoring of each component 0 score indicates (normal) , 1 score indicates (mild abnormality) and 2 scores indicate (sever abnormality). Total score (0-3) indicates minimal risk of post-extubation complications ,4-6 indicates moderate risk of complications and 7-10 indicates high risk of post-extubation complications.
change from the baseline in swallowing on Pediatric Dysphagia Screening Questionnaire (PDSQ) | The first measurement time will be From extubation of mechanical ventilation up to 1 week"7 th day's post-extubation". The second time will be from extubation up to 2 week"14th day's" post-extubation
  it designed to identify children at risk for oropharyngeal dysphagia. scoring of each component 0 score indicates (no difficultly) ,1 score indicates (mild difficulty)2 scores (moderate difficulty) and 3 score indicates (severe difficulty). Total score (0-5) indicates minimal or to no dysphagia risk ,6-10 indicates to some dysphagia risk, 11-15 indicates high dysphagia risk and 16-18 indicates Severe dysphagia risk.
change from baseline of normal oral intake of the children on the Pediatric Functional Oral Intake Scale (P-FOIS) | The first measurement time will be From extubation of mechanical ventilation up to 1 week"7 th day's post-extubation". The second time will be from extubation up to 2 week"14th day's" post-extubation
  it includes a 6-point scale used to assess a child's oral intake ability. It categorizes intake into seven levels, ranging from complete dependence on non-oral feeding to successful oral intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr Ash Shaykh, Kafr el-Sheikh, Egypt,, Egypt

IPD SHARING:
Plan to Share IPD: No